CLINICAL TRIAL: NCT06207396
Title: Characteristics of Spiking in Ghent: A Multicentric Prospective Observational Study
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2023-0004
Record Dates: First submitted 2023-12-05; First posted 2024-01-17 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Intoxication; Unintended Ingestion of Product
MeSH Terms: interventions — Urinalysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and/or urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serum and urine analysis — Spiking will be analyzed by immunoassay testing and high-resolution screening

SUMMARY:
This study aims to document the incidence and characteristics of spiking in the Ghent region, both anamnestically and by toxicological analysis.

Spiking will be analyzed by immunoassay testing and high-resolution screening according to the protocol in the laboratory of UZ Gent;

DETAILED DESCRIPTION:
This study aims at objectivating and characterizing the patients with alleged spiking in the city of Ghent.

Every patient who presents at one of the four (out of four) emergency departments of Ghent, with a suspicion of spiking (drink/food/needle-spiking included), will be offered to take part of this study.

The study entails a list of questions for the patient regarding demographics, recent own medication/drug/alcohol use and experienced symptoms; whilst the caregiver (doctor/nurse) completes a questionnaire regarding symptoms at time of presentation.

For a presentation within 48h after event, both blood and urine samples are requested from the patient. When presenting between 48h and 96h after the event, only urine samples are requested.

On this samples, IA and LC-GCMS according to the UNODOC standards ("Guidelines for the Forensic analysis of drugs facilitating sexual assault and other criminal acts") to objectify exogenous products.

On request of the patient, these results can be added to the medical file of the patient.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Patient self-reports suspicion of spiking OR there is a suspicion of spiking by physician, police, paramedics or patient's companions
* willingness to provide urine and/or blood samples (depending on timing after event)

Exclusion Criteria:

* Reporting more than 5 days after spiking
* Unable to reliably complete the questionnaire (can be after clinical observation/recovery).
* Not declaring proficiency in the language in which informed consent is offered (Dutch/English).
* Not agreeing to the informed consent.
* Do not consent to blood and urine collection and/or analysis.
* There is a suspicion of Drug Facilitated Sexual Assault (to be referred to Care Center Sexual Violence, ZSG, where parallel study is ongoing).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult population (18+, all genders) presenting with alleged spiking to the emergency department
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
What is the incidence of spiking in adult patients presenting to the emergency departments of the four Ghent hospitals with suspected spiking? | 19 months
  Number of patients presenting to the ED with spiking
What is the type of product and mode of administration used in spiking | 19 months
  Defining type of products and mode of administration
What are patient characteristics of patients with spiking | 19 months
  Demographic features of the patients diagnosed with spiking
In what type of places does spiking occur in Ghent | 19 months
  Location of spiking event

CONTACTS AND LOCATIONS:
Locations (4):
- Belgium (4):
  - AZ Maria Middelares, Ghent
  - Spoedgevallendienst AZ Jan Palfijn, Ghent
  - Spoedgevallendienst AZ St. Lucas, Ghent
  - Spoedgevallendienst, Ghent